CLINICAL TRIAL: NCT05808426
Title: Randomized Trial of Online Mahjong Intervention to Promote Cognitive Function and Health Status in Community-dwelling Middle Aged and Older Adults.
Brief Title: Benefits of Online Mahjong by Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: YM108123F_M
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2020-06

CONDITIONS: Aged
Keywords: online Mahjong; physical activity; cognitive function; quality of life in older adults
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: This study is a single-blind, parallel-group randomized controlled trial. Eligible participants were allocated randomly 1:1, without stratification, to either the intervention or the control group, according to a computer-generated random number sequence.
Who Masked: Investigator
Masking Description: Participants were not explicitly informed about their group assignment and there was no contact between study investigators and participants during the study period. The intervention allocation was masked from investigators by anonymized coding, and the individuals who were assigned interventions were not involved in assessing outcomes and analyzing data. The investigators also avoided any potential interactions between participants in either intervention group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- observation with no intervention group (No Intervention): The control group only performed routine data collection; the research assistant asked the subjects about their usual activities by telephone every month to understand their physical activity in this half of the year.
- Mahjong group (Experimental): The experimental group intervened a Bonus Winner Mahjong developed by Bonus Winner Online Entertainment Co., Ltd. The participants in experimental group played three times a week, each time requiring at least lasting 30 minutes, for half of a year.
  Interventions: Device: Bonus Winner Mahjong

INTERVENTIONS:
Device: Bonus Winner Mahjong — Bonus Winner Mahjong developed by Bonus Winner Online Entertainment Co., Ltd. The participants in experimental group played three times a week, each time requiring at least lasting 30 minutes, for half of a year.
  Arms: Mahjong group

SUMMARY:
This study aims to examine the clinical efficacy of online Mahjong in improving physical health, cognitive performance, happiness, laboratory biomarkers, and structural brain imaging (magnetic resonance imaging, MRI) by a randomized controlled trial design, and hopefully to expand the scope of healthy aging intervention activities with strong scientific evidence.

DETAILED DESCRIPTION:
Psychomotor function among older adult's decline was associated with reducing people interaction during pandemic has been reported. The research focused on examining the benefit and efficacy of digital based Mahjong games with 6-month intervention is very limited or none. A random control design was conducted with comparing intervention group and with control group, followed the CONSORT guidelines. Six months program was intervened to ensure the impact of the intervention. Primary outcome is brain imagery changes between groups, which showed changes in temporal fusiform cortex but not in resting-state fMRI. The total score of MoCA, delayed recall was increase from baseline to after intervention in experimental group. Overall cognitive function and visuospatial/executive, in experimental group improved more than control group. Improving self-rating daily health status as associated with achievement rate of Mahjong game. Increasing level of resilience was associated with demoralization level, subtraction of cognitive function, and 5th month walking steps. In addition, affecting incased self -rate overall heath was related to demoralization. In short, online mahjong intervention has positive impact on older adults in cognitive function , resilience, demoralization and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 55 years old.
2. More than 6 years of formal education.
3. Can communicate in Mandarin and Taiwanese.
4. Can accept MRI examination without claustrophobia.
5. Can understand the research process, meet the requirements of the research, and can sign the consent form and participate in the subject.

Exclusion Criteria:

1. Have engaged in any Mahjong games in the past three months.
2. Engaged in Mahjong games more than three times per year in the past three years.

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Change in MRI study from baseline to 6 months in the intervention group. | baseline and 6 months
  Change in MRI study from baseline to 6 months in the intervention group.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | baseline and 6 months
  Cognitive function measure by MoCA , which comprise a 30-question test.Score range: 0-30, and a score of 26 and higher is considered normal.
EuroQol instrument (EQ-5D) | baseline and 6 months
  Quality of life measure by EQ-5D, which include five questions on mobility, self care, pain, usual activities, and psychological status. Score range: There are three level of the answers for each question, the maximum score of 1 refers to the best condition without problem, and higher scores refers more severe of the issue. Moreover, the visual analogue scale (VAS) which from 0-100, higher score indicating better health status.
International Physical Activity Questionnaire (IPAQ) | baseline and 6 months
  Physical activity measured by IPAQ, indicates that spent being physically active within the prior 7 days. Score range: There are no established thresholds for presenting MET-minutes, the IPAQ Research Committee proposes that reported as comparisons of median values and interquartile ranges for different populations.
Brief Resilience Scale (BRS) | baseline and 6 months
  Resilience measured by BRS to assess ability to bounce back or recover from stress and adversity. Score range: 6-30, and higher scores refers to higher level of resilience.
Demoralization Scale-Mandarin Version (DS-MV) | baseline and 6 months
  Demoralization measure by DS-MV, comprised 24 items and each rated on a five-point Likert scale.Score range: 0-96, and cut-off point score ≥30 was considered to identified demoralization.

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Kung Chen, PhD, Principal Investigator — Center for Healthy Longevity and Aging Sciences,National Yang Ming Chiao Tung University
Locations (1):
- Center for Geriatrics and Gerontology, Taipei Veterans General Hospital, Taipei, Taiwan